CLINICAL TRIAL: NCT01022164
Title: Safety and Efficacy in the Use of Fibrin Glue in Vitreoretinal Surgery
Brief Title: Use of Fibrin Glue in Vitreoretinalsurgery
Acronym: fibringlue
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Undefined
Sponsor: Asociación para Evitar la Ceguera en México (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: APEC0005
Record Dates: First submitted 2009-11-29; First posted 2009-12-01 (Estimated); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Surgery
Keywords: fibrin glue; vitrectomy; safety and efficacy of fibrin glue
MeSH Terms: interventions — Fibrin Tissue Adhesive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- fibrin glue (Other)
  Interventions: Procedure: fibrin glue

INTERVENTIONS:
Procedure: fibrin glue
  Other Names: Beriplast

SUMMARY:
To study the Safety and Efficacy of the use of fibrin glue in vitreoretinal surgery

ELIGIBILITY:
Inclusion Criteria:

* Vitreorretinal procedures that require suture

Exclusion Criteria:

* None

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-05 (Actual); Primary Completion 2009-11 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Asociacion para Evitar la Ceguera en Mexico, México, Mexico